CLINICAL TRIAL: NCT01324557
Title: Insulin Pump Therapy and Continuous Glucose Monitoring in Diabetic Continuous Ambulatory Peritoneal Dialysis (CAPD) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Division fo Nephrology, Guangdong General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InsulinPump
Record Dates: First submitted 2011-03-09; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes; Poor Glycemic Control
Keywords: Continuous glucose monitoring; CAPD patients; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSII (Experimental): Optimized subcutaneous insulin infusion by means of continuous subcutaneous insulin infusion (CSII)
  Interventions: Procedure: CSII and MDI
- MDI (No Intervention): MDI: Control Optimized subcutaneous insulin by multiple daily injections (MDI)
  Interventions: Procedure: CSII and MDI

INTERVENTIONS:
Procedure: CSII and MDI — The aims of this study are to assess the potential efficacy and safety of insulin pump(MiniMed Paradigm® REAL-Time Revel™ Insulin Pump) to improve glycemic control in conjunction with continuous glucose monitoring (CGMS) for diabetic CAPD Patients.

SUMMARY:
The aims of this study are to assess the potential efficacy and safety of insulin pump to improve glycemic control in conjunction with continuous glucose monitoring (CGMS) for diabetic continuous ambulatory peritoneal dialysis (CAPD) patients.

DETAILED DESCRIPTION:
Diabetic nephropathy now accounts for 20% to 40% of all patients entering end-stage renal failure (ESRF) programs. The quality of glycemic control is known to be an important determinant of the rate of progression of patients with diabetic continuous ambulatory peritoneal dialysis (CAPD) patients. Diabetic CAPD patients are usually treated with dialysis fluids utilizing glucose as the osmotic agent to provide ultrafiltration. Most of diabetic CAPD patients had HbA1c readings above 7% despite the recommendation to keep the reading below 7%.

The continuous blood glucose monitor (CGMS) has recently offered an opportunity to monitor blood glucose at 5-minute intervals for 72 continuous hours in diabetic patients. The CGMS patterns reveal blood glucose tracings well above the recommended standards of control in most of the diabetic CAPD patients.

Good glycemic control is often difficult to maintain in diabetic patients treated with CAPD because they are continuously exposed to high concentrations of glucose in peritoneal dialysate. However, recent studies have suggested that diabetic patients who use insulin pump has been shown to reduce glycated hemoglobin levels without an increased risk of hypoglycemia, as compared with a regimen of multiple daily insulin injections, but results in diabetic CAPD patients have not been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 70 years old at registration
2. Type 1 or Type 2 Diabetic CAPD patients for at least 3 month and less than 60 months
3. Hemoglobin A1c of at least 7.5% at registration Kt/V is greater than 1.7

Exclusion Criteria:

1. Have peritonitis in recent 3 months other active bacterial infections
2. Unstable clinical conditions or evidence of malignancy
3. Pregnancy
4. Non-diabetic ESRD patients
5. Individuals already receiving diabetes therapy via an insulin pump

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) measurement | 24 week follow-up

SECONDARY OUTCOMES:
The frequency of hypoglycemic episodes | at 24 week follow-up
  Glycemic control, Glycosylated hemoglobin (HbA1c) measurement; Frequency of adverse events; Frequency of clinically significant abnormal laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Shi Wei, PHD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China